CLINICAL TRIAL: NCT06703684
Title: TCM Syndrome Differentiation of Type 2 Diabetes Comorbid With Metabolic Syndrome
Brief Title: TCM Syndrome Differentiation of T2DM & MetS
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZHANG Jialing, Principal Investigator, Hong Kong Baptist University
Other Study IDs: REC/23-24/0564
Record Dates: First submitted 2024-11-17; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cross-sectional observational study — This is a cross-sectional observational study. No intervention will be given.

SUMMARY:
This study aims to include type 2 diabetes (T2DM) patients comorbid with metabolic syndrome (MetS). The primary aim of the study is to investigate the TCM (Traditional Chinese Medicine) syndrome differentiation of T2DM comorbid with MetS.

DETAILED DESCRIPTION:
This study adopts a cross-sectional design, to include type 2 diabetes (T2DM) patients comorbid with metabolic syndrome (MetS). The primary aim of the study is to investigate the TCM (Traditional Chinese Medicine) syndrome differentiation of patients with T2DM and MetS. The demographic data, anthropometric data, fasting glucose and HbA1c, lipid panel, TCM syndrome differentiation information, dietary assessment, physical activity, sleep quality, and quality of life, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age between 18-75y.
* (2) Diagnosed with Type 2 diabetes.
* (3) Diagnosed with Metabolic Syndrome according to Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition) from Chinese Diabetes Society. People who meet 3 of the following diagnostic criteria or more can be diagnosed as Metabolic Syndrome: (a) Abdominal obesity: waist circumference ≥ 90cm for male and ≥ 85cm for female; (b) Hyperglycemia: Fasting blood glucose ≥ 6.1mmol/L or 2-hour postprandial glucose ≥ 7.8mmol/L and/or those who have been diagnosed with hyperglycemia and in treatment; (c) Hypertension: blood pressure ≥ 130/85mmHg and/or those who have been diagnosed with hypertension and in treatment; (d) Fasting triglyceride ≥ 1.70mmol/L; (e) Fasting HDL-C < 1.04mmol/L.
* (4) Clearly understand the content of the study and voluntarily sign the informed consent form.
* (5) Provide complete data (basic information, TCM diagnosis data, and blood test results).

Exclusion Criteria:

* (1) Diagnosed with type 1 diabetes, steroid-induced diabetes, gestational diabetes, or specific types of diabetes.
* (2) Diabetes accompanied by severe complications such as diabetic nephropathy, diabetic ketoacidosis, etc.
* (3) Secondary obesity (e.g., secondary to pituitary inflammation, tumor, etc.).
* (4) Secondary hypertension (e.g., pheochromocytoma, renal hypertension, etc.).
* (5) Secondary hyperlipidemia (e.g., hypothyroidism, nephrotic syndrome, etc.).
* (6) With severe heart, liver, or kidney disease or bleeding disorders, or with other serious diseases (e.g. cancer, dementia, etc.).
* (7) With severe mental disorders, speech or hearing impairments.
* (8) Pregnancy or lactation female.
* (9) Currently join other clinical trial.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study adopts a cross-sectional design, to include subjects with type 2 diabetes (T2DM) patients comorbid with metabolic syndrome (MetS), irrespective of T2DM duration.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TCM syndrome differentiation | Baseline
  A registered Chinese medicine practitioner (CMP) will conduct the TCM syndrome differentiation assessment using a standardized questionnaire, incorporating four TCM diagnostic methods.

SECONDARY OUTCOMES:
Demographic data | Baseline
  Gender, date of birth, living status, marital status, education level, income status, occupation, work status, smoking history, alcohol consumption history, allergy history, medical history, etc.
Anthropometric data | Baseline
  Anthropometric measurements such as skin fold thickness measurements.
Fasting glucose | Baseline
  Fasting glucose level is measured.
Lipid panel | Baseline
  Total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein levels are measured.
Hemoglobin A1c (HbA1c) | Baseline
  HbA1C level is measured.
Framingham Stroke Risk Score (FSRS) | Baseline
  Framingham Stroke Risk Score (FSRS) is calculated based on variables such as age, cholesterol, blood pressure, diabetes, and smoking. Individuals with low risk have 10% or less risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | Baseline
  International Physical Activity Questionnaire Short Form (IPAQ-SF) has been recommended as a cost-effective method to assess physical activity. The IPAQ-SF evaluates the number of days and time spent performing MVPA, walking, and sitting in bouts of at least 10 min over the previous 7 days. The summary score is expressed in PA metabolic equivalent of task (MET)-min per day or week.
Audit of diabetes-dependent quality of Life (ADDQoL) | Baseline
  Audit of diabetes-dependent quality of Life (ADDQoL) consists of 2 overview items; one measures generic overall QoL and a further 19 items are concerned with the impact of diabetes on specific aspects of life. The scales range from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Lower scores reflect poorer QOL.
Pittsburgh sleep quality index (PSQI) | Baseline
  Pittsburgh sleep quality index (PSQI) was a 19-item questionnaire used to assess sleep dysfunction over a 1-month period. The total score for the PSQI varies from 0 to 21. A PSQI total score >5 is indicative of poor sleep.
Dietary assessment | Baseline
  Dietary intake will be assessed via food frequency questionnaire (FFQ). The 60-item FFQ (<30 min for administration) with food items will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jialing ZHANG, PhD, Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang J, Wong HK, Lin Z, Zhong S, Ma M, Wang X. Traditional Chinese Medicine Syndrome Differentiation of Adult Patients With Type 2 Diabetes and Metabolic Syndrome: Protocol for a Cross-Sectional Study. JMIR Res Protoc. 2026 Jan 23;15:e86217. doi: 10.2196/86217. PMID 41576380